CLINICAL TRIAL: NCT05352919
Title: A Multicenter, Randomized, Dose-Blind, Phase 3 Long-Term Extension Study to Evaluate Continuous Safety and Efficacy of Litifilimab (BIIB059) in Adult Participants With Active Systemic Lupus Erythematosus
Brief Title: An Extension Study to Learn More About the Long-Term Safety of Litifilimab (BIIB059) Injections and Whether They Can Improve Symptoms of Adult Participants Who Have Systemic Lupus Erythematosus
Acronym: EMERALD
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 230LE306; 2021-006378-22 (EudraCT Number); 2023-505635-13 (Other: EU CTIS Number)
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Lupus Erythematosus; Systemic Autoimmune Diseases; Connective Tissue Diseases; Immune System Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Connective Tissue Diseases; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Litifilimab Low Dose (Experimental): Participants who are receiving background nonbiologic lupus standard of care (SOC) therapy and received litifilimab low dose, subcutaneously (SC), every 4 weeks (Q4W) during the parent Phase 3 studies (i.e. studies 230LE303 [NCT04895241] or 230LE304 [NCT04961567]) will continue to receive litifilimab low dose, SC, Q4W from Day 1 up to 152 weeks with an additional dose of litifilimab-matching placebo at Week 2.
  Participants who are receiving background nonbiologic lupus SOC therapy and received litifilimab-matching placebo in the parent Phase 3 studies (i.e. studies 230LE303 [NCT04895241] or 230LE304 [NCT04961567]) will be randomized to receive litifilimab low dose, SC, Q4W from Day 1 up to 152 weeks with an additional dose at Week 2.
  Interventions: Drug: Litifilimab; Drug: Litifilimab-matching placebo
- Litifilimab High Dose (Experimental): Participants who are receiving background nonbiologic lupus SOC therapy and received litifilimab high dose, SC, Q4W during the parent Phase 3 studies (i.e. studies 230LE303 [NCT04895241] or 230LE304 [NCT04961567]) will continue to receive litifilimab high dose, SC, Q4W from Day 1 up to 152 weeks with an additional dose of litifilimab-matching placebo at Week 2.
  Participants who are receiving background nonbiologic lupus SOC therapy and received litifilimab-matching placebo in the parent Phase 3 studies (i.e. studies 230LE303 [NCT04895241] or 230LE304 [NCT04961567]) will be randomized to receive litifilimab high dose, SC, Q4W from Day 1 up to 152 weeks with an additional dose at Week 2.
  Interventions: Drug: Litifilimab; Drug: Litifilimab-matching placebo

INTERVENTIONS:
Drug: Litifilimab — Administered as specified in the treatment arm.
  Other Names: BIIB059
Drug: Litifilimab-matching placebo — Administered as specified in the treatment arm.
  Other Names: BIIB059

SUMMARY:
In this study, researchers will learn more about a study drug called litifilimab (BIIB059) in participants with systemic lupus erythematosus (SLE). The study will focus on participants who have active disease and are already taking standard of care medications. These may include antimalarials, steroids, and immunosuppressants. This is an extension study of 230LE303 and 230LE304 (TOPAZ-1 and TOPAZ-2). It will enroll participants who completed the treatment periods of either one of the parent studies.

The main objective of the study is to learn more about the long-term safety of litifilimab. The main question researchers want to answer is:

- How many participants have adverse events and serious adverse events? Researchers will also learn about the effect litifilimab has on controlling symptoms of SLE and lowering its activity. They will measure symptoms of SLE over time using a variety of scoring tools. These include the SLE Responder Index (SRI), the Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K), and the British Isles Lupus Activity Group-2004 (BILAG-2004), among others.

Researchers will also study how participants' immune systems respond to litifilimab. Additionally, they will measure the effect litifilimab and SLE have on the quality of life of participants using a group of questionnaires.

The study will be done as follows:

* The Week 52 visit of studies 230LE303 and 230LE304 will be Day 1 of this study.
* Participants who were receiving either a high or low dose of litifilimab in the parent studies will continue receiving the same doses.
* Participants who were receiving placebo in the parent studies will be randomized to receive either a high or low dose of litifilimab.
* All participants will receive litifilimab as injections under the skin once every 4 weeks. The treatment period will last 156 weeks. Participants may continue to take their standard of care medications.
* Neither the researchers nor the participants will know which doses of litifilimab the participants are receiving.
* There will be a follow-up safety period that lasts up to 24 weeks.
* In total, participants will have up to 47 study visits. The total study duration for participants will be up to 180 weeks.

Optional Substudy: Some participants may be invited to join an optional substudy after being in the main study for at least 4 months. This substudy will test a new injector device for giving litifilimab. The injector device is an automatic device that delivers the full dose in one injection without needing to push a plunger. Researchers will compare the safety and tolerability of the injector device and how the body reacts to it to the current prefilled syringe method. The substudy will last 3 months and will include about 120 participants.

DETAILED DESCRIPTION:
This is an extension study for all participants who completed study 230LE303 (NCT04895241) and 230LE304 (NCT04961567) (parent phase 3 studies) through Week 52 and did not discontinue litifilimab or placebo. Eligible participants from parent phase 3 studies will be followed for up to 180 weeks.

The primary objective of this study is to evaluate the long-term safety and tolerability of litifilimab in participants with active systemic lupus erythematosus (SLE).

The secondary objectives of this study are to evaluate the long-term effect of litifilimab on disease activity in participants with SLE, to evaluate the long-term effect of litifilimab in participants with SLE in maintaining low disease activity, to evaluate the effect of litifilimab in participants with active SLE in preventing irreversible organ damage, to assess long-term use of oral corticosteroid (OCS) with participants receiving litifilimab treatment, to assess the impact of litifilimab on participant-reported Health-Related Quality-of-Life Questionnaire (HRQoL), symptoms, and impacts of SLE, to evaluate long-term effect of litifilimab on laboratory parameters, and to evaluate immunogenicity of litifilimab.

A phase-3, randomized, dose-blind, substudy is added in this extension study for all participants who have been enrolled in the 230LE306 Phase 3 LTE study for a minimum of 4 months and have at least four remaining visits in the Phase 3 LTE study.

The primary objective of this substudy is to evaluate the safety of injector device used for administering litifilimab in participants with active SLE.

The secondary objective of this substudy is to evaluate the tolerability of injector device used for administering litifilimab in participants with active SLE.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who completed 1 of the 52-week of the double-blind placebo-controlled, parent Phase 3 studies (230LE303 (NCT04895241) and 230LE304 (NCT04961567)) on study treatments with either litifilimab or placebo to Week 48 and attended the last study assessment visit at Week 52.

Key Exclusion Criteria:

* Early parent Phase 3 studies treatment terminators (participants who discontinued study treatment before Week 52)
* Early parent Phase 3 studies terminators (participants who withdrew from study participation and did not complete the 52-week treatment period)
* Participants who developed moderate-to-severe worsening of organ-specific lupus manifestations that would require a change in antimalarials and/or immunosuppressive therapy (initiation of new treatment or increase in dose above the allowed maximum dose)
* Use of other investigational drugs or off-label drugs used to treat SLE, cutaneous lupus, or lupus nephritis during the parent Phase 3 studies.

NOTE: Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2030-03-29 (Estimated); Study Completion 2030-03-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to Week 180
  An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is an AE that started or worsened in severity after the first dose of study treatment through 28 days after the last dose of study treatment or end of study (EOS) date, whichever comes earlier.
Number of Participants with Serious Adverse Events (SAEs) | Up to Week 180
  An SAE is any untoward medical occurrence that at any dose results in death, in the view of the Investigator, places the participant at immediate risk of death (a life threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, and is a medically important event.

SECONDARY OUTCOMES:
Percentage of Participants who Achieved an Systemic Lupus Erythematosus Responder Index (SRI)-4 Response | Up to Week 180
  SRI-4 is a composite endpoint defined as the following:
  * A reduction from baseline of ≥4 points in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI-2K) score.
  * No new organ system affected, as defined by no new British Isles Lupus Activity Group-2004 (BILAG-2004 grade A) and no more than 1 new BILAG 2004 grade B versus previous visit.
  * No worsening from baseline in lupus disease activity as defined by <0.3-point increase on 3-point Physician's Global Assessment (PGA) visual analog scale (VAS).
  * No violation of protocol-specified medication rules
Percentage of Participants With at Least 4 Joints (Both Swollen and Tender) at Baseline who Achieved a Joint-50 Response | Up to Week 180
  Joint-50 response is a 50% reduction in total active joint count from baseline. An active joint is defined as a joint with pain and signs of inflammation (e.g., tenderness, swelling or effusion). A 28-joint assessment will be performed to determine the active joint count, which is defined as the sum of tender and swollen joint counts.
Percentage of Participants With a Cutaneous Lupus Erythematosus Disease Area and Severity Index - Activity (CLASI-A) Score ≥10 at Baseline who Achieved a CLASI-50, CLASI-70, and CLASI-90 Response | Up to Week 180
  CLASI score is used to evaluate lupus skin manifestations. The activity scale (CLASI-A) includes measurements of erythema, scale and hypertrophy, and mucous membrane disease. Each part of the body is listed separately, from the scalp to the feet, in addition to sections focusing on mucous membrane involvement and alopecia. Points are given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. Scores for each area are assigned based on the most severe lesion within the area of interest. CLASI-A scores of 0 to 9, 10 to 20, and 21 to 70 represent disease severity of mild, moderate, and severe, respectively. CLASI-50, CLASI-70, and CLASI-90 responders are defined as ≥ 50%, ≥ 70%, and ≥ 90% improvement in CLASI-A score from baseline at the specified timepoint.
Percentage of Participants who Achieved a British Isles Lupus Assessment Group based Composite Lupus Assessment (BICLA) Response | Up to Week 180
  BICLA is a composite endpoint defined as the following:
  * BILAG-2004 improvement, defined as all of BILAG-2004 Grade A at baseline improved to B, C, or D and all of BILAG-2004 Grade B at baseline improved to C or D.
  * No BILAG-2004 worsening in other BILAG-2004 organ systems such that there are no new BILAG-2004 Grade A or greater than 1 new BILAG-2004 Grade B.
  * No worsening in the SLEDAI-2K total score compared to baseline.
  * No worsening from baseline in lupus disease activity as defined by <0.3-point increase on 3-point PGA VAS.
  * No violation of protocol-specified medication rules.
Annualized Severe Safety of Estrogens in Systemic Lupus Erythematosus National Assessment - Systemic Lupus Erythematosus Disease Activity Index Flare Index (SFI) Flare Rate | Up to Week 156
  A severe flare is defined as any of the following:
  * Change in SLEDAI instrument score to >12
  * New or worse: central nervous system SLE; vasculitis; nephritis; myositis; platelets <60,000/mL, or hemolytic anemia with hemoglobin <7 grams per deciliter (g/dL) or decrease in hemoglobin >3 g/dL and requiring: doubling prednisone dose, increase to >0.5 milligrams per kilograms per day (mg/kg/day) or hospitalization
  * Increase in prednisone dose to >0.5 mg/kg/day
  * New requirement for cyclophosphamide, azathioprine, methotrexate, or mycophenolate for SLE activity
  * Hospitalization for SLE activity
  * Increase in PGA score to >2.5
Percentage of Time Spent in Lupus Low Disease Activity State (LLDAS) | Up to Week 180
  LLDAS is a composite endpoint defined as the following:
  i. SLEDAI-2K score ≤ 4, with no activity in a major organ system (renal, central nervous system, cardiopulmonary, vasculitis, fever); and ii. No new features of lupus disease activity compared with the previous assessment; and iii. SELENA-SLEDAI PGA ≤ 1; and iv. Current prednisone (or equivalent) dose ≤ 7.5 mg/day; and v. Standard maintenance doses of immunosuppressive drugs and approved biological agents.
  "No new features" is defined as any new SLEDAI-2K component that was not present at the previous assessment. The SELENA-SLEDAI PGA Scale ranges from 0-3, where 0 is no disease activity and 3 is maximum disease activity. "Standard maintenance doses" include drugs limited to those allowed per protocol.
Percentage of Participants With Sustained LLDAS | Up to Week 180
  LLDAS is a composite endpoint defined as the following:
  i. SLEDAI-2K score ≤ 4, with no activity in a major organ system (renal, central nervous system, cardiopulmonary, vasculitis, fever); and ii. No new features of lupus disease activity compared with the previous assessment; and iii. SELENA-SLEDAI PGA ≤ 1; and iv. Current prednisone (or equivalent) dose ≤ 7.5 mg/day; and v. Standard maintenance doses of immunosuppressive drugs and approved biological agents.
  "No new features" is defined as any new SLEDAI-2K component that was not present at the previous assessment. The SELENA-SLEDAI PGA Scale ranges from 0-3, where 0 is no disease activity and 3 is maximum disease activity. "Standard maintenance doses" include drugs limited to those allowed per protocol.
Duration of Sustained LLDAS as Defined by the Number of Visits in LLDAS | Up to Week 180
  LLDAS is a composite endpoint defined as the following:
  i. SLEDAI-2K score ≤ 4, with no activity in a major organ system (renal, central nervous system, cardiopulmonary, vasculitis, fever); and ii. No new features of lupus disease activity compared with the previous assessment; and iii. SELENA-SLEDAI PGA ≤ 1; and iv. Current prednisone (or equivalent) dose ≤ 7.5 mg/day; and v. Standard maintenance doses of immunosuppressive drugs and approved biological agents.
  "No new features" is defined as any new SLEDAI-2K component that was not present at the previous assessment. The SELENA-SLEDAI PGA Scale ranges from 0-3, where 0 is no disease activity and 3 is maximum disease activity. "Standard maintenance doses" include drugs limited to those allowed per protocol.
Annual Change From Baseline Value From the Parent Phase 3 Studies in Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index (SDI) Score | Up to Week 156
  SDI score is used to assess the accumulated damage in participants with SLE. It assess 12 organ systems and records damage in participants with lupus, regardless of its cause. Damage could be due to previous disease activity, medication, or intercurrent illness (such as surgery or cancer). To distinguish between active inflammation and damage, an item must be present for at least 6 months. It is assumed that persistent inflammation (for at least 6 months) would result in tissue injury and hence damage. SDI is evaluated on a scale 0-47 with higher score indicating higher damage.
Cumulative Exposure to OCS Over Time | Up to Week 156
Percentage of Participants With OCS ≤7.5 mg | Up to Week 156
Percentage of Participants With OCS ≤5 mg | Up to Week 156
Change From Baseline in Lupus-Specific Health-Related Quality-Of-Life (LupusQoL) Score | Up to Week 156
  The LupusQoL is a participant-reported, lupus-specific, HRQoL questionnaire consisting of 34 items grouped in 8 domains: physical health, pain, planning, intimate relationships, burden to others, emotional health, body image and fatigue. Participants indicate their responses on a 5-point Likert response format, where 4 = never, 3 = occasionally, 2 = a good bit of the time, 1 = most of the time, and 0 = all the time. A LupusQoL score for each domain will be reported on a 0 to 100 scale, with greater values indicating better HRQoL.
Change From Baseline in Short Form Health Survey-36 (SF-36) (Acute Version) Score | Up to Week 156
  The SF-36 is a 36-item scale which assesses HRQoL in 8 domains: limitations in physical activities due to health problems, limitations in social activities due to physical or emotional problems, limitations in usual role activities due to physical health problems, bodily pain, general mental health (psychological distress and well-being), limitations in usual role activities due to emotional problems, vitality (energy and fatigue), general health perceptions. The SF-36 (Acute Version) form asks for participants to reply to questions (items) according to how they have felt over a specifically defined period of time. Items 1-4 primarily contribute to the physical component summary (PCS) score of the SF-36. Items 5-8 primarily contribute to the mental component summary (MCS) score of the SF-36 where higher scores indicate best health. Scores on each item are summed and averaged (range: 0=worse health to 100=best possible health).
Change From Baseline in European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3L) | Up to Week 156
  The EQ-5D is a standardized generic measure of health status developed by the European Quality of Life Group. This study uses the EQ-5D-3L version of the instrument. This instrument consists of 2 sections. The first section comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. All dimensions are measured on a 3-point scale, 1: No problems; 2: Some problems; 3: Extreme problems. The second section comprises the Visual Analogue Scale, which records the respondent's self-rated health on a vertical scale ranging from 0 to 100, lower scores indicate the worst possible health state.
Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score | Up to Week 156
  The FACIT-Fatigue is a participant-administered HRQoL questionnaire that evaluates participant's fatigue in 5 broad categories: physical well-being, social/family well-being, emotional well-being, functional well-being and additional concerns. The level of fatigue is measured by questions assessed on a 5-point scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much). The responses for each item are added to obtain a total score which ranges from 0 to 52, with a higher score indicating less fatigue.
Change From Baseline in Patient Health Questionnaire-9 (PHQ-9) Score | Up to Week 156
  The PHQ-9 is a participant-administered HRQoL questionnaire to screen for the presence and severity of depression. The PHQ-9 is a participant-reported outcome (PRO) that is used to measure depression in adults. It contains 9 questions, with a 2 week recall period. The PHQ-9 yields an overall severity score that can range from 0 to 27 with the following severity scores: 0-4 = none; 5-9 = mild; 10-14 = moderate; 15-19 = moderate-to-severe; and 20-27 = severe.
Change From Baseline in Work Productivity and Activity Impairment (WPAI):Lupus Score | Up to Week 156
  WPAI questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. Each score ranges from 0 to 100, with higher numbers indicating greater impairment and less productivity.
Change from Baseline in Patient Global Assessment (PtGA) Score | Up to Week 156
  The PtGA is participant-administered, single-item question evaluating the impact of health and illness, with responses ranging from very poor to very well on a 100 mm VAS. The participant will consider the previous week when addressing this question.
Number of Participants with Clinically Relevant Abnormalities in Standard Laboratory Parameters | Up to Week 180
  Standard laboratory parameters will include hematology, blood chemistry, urinalysis, and coagulation.
Number of Participants with Clinically Relevant Abnormalities in Electrocardiogram (ECG) Results | Up to Week 156
Number of Participants with Antibodies to Litifilimab | Up to Week 180

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (179):
- United States (36):
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - Wallace Rheumatic Study Center, Beverly Hills, California
  - Care Access Research - Huntington Beach, Huntington Beach, California
  - Providence Facey Medical Foundation, Mission Hills, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - University of Colorado Denver, Aurora, Colorado
  - Georgetown University Hospital-Medstar, Washington D.C., District of Columbia
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - Highlands Research Institute, Avon Park, Florida
  - Clinical Research of West Florida - Corporate, Clearwater, Florida
  - GNP Research at Mark Jaffe, MD, Cooper City, Florida
  - Omega Research Consultants, DeBary, Florida
  - Life Clinical Trials, Margate, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - AdventHealth Medical Group, Tampa, Florida
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - AA MRC LLC Ahmed Arif Medical Research Center, Flint, Michigan
  - Precision Comprehensive Clinical Research Solutions, Rochester Hills, Michigan
  - Saint Louis Rheumatology, St Louis, Missouri
  - NYU Langone Brooklyn, Brooklyn, New York
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - West Tennessee Research Institute, Jackson, Tennessee
  - Ramesh C Gupta, MD, Memphis, Tennessee
  - Arthritis & Rheumatology Research Institute, Allen, Texas
  - Tekton Research - PARENT, Austin, Texas
  - Accurate Clinical Research, Baytown, Texas
  - Precision Comprehensive Clinical Research Solution, Colleyville, Texas
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Accurate Clinical Research, Inc., Humble, Texas
  - R and H Clinical Research, Katy, Texas
  - Sun Research Institute, LLC, San Antonio, Texas
  - Advanced Rheumatology of Houston, The Woodlands, Texas
  - Swedish Medical Center, Seattle, Washington
- Argentina (16):
  - Organizacion Medica de Investigacion (OMI), CABA, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Policlìnica Red Omip S.A - Ensayos Clinicos GC, Mar del Plata, Buenos Aires
  - Centro Dermatologico Schejtman, San Miguel, Buenos Aires
  - Centro Medico Barrio Parque, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Instituto CAICI, Rosario, Santa Fe Province
  - Clinica Mayo de Urgencias Medicas Cruz Blanca SRL, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Hospital Italiano de La Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Buenos Aires
  - Centro Medico Dra Laura Maffei Investigacion Clinica Aplicada, Ciudad Autonoma Buenos Aires
  - STAT Research S.A., Ciudad Autonoma Buenos Aires
  - Sanatorio Allende, Córdoba
  - Instituto de Reumatologia, Mendoza
  - CER San Juan Centro Polivalente de Asistencia e Inv. Clinica, San Juan
- Centre Hospitalier Universitaire de Liege, Liège, Belgium
- Brazil (16):
  - HUWC - UFC - Hospital Universitário Walter Cantídio - Universidade Federal do Ceará, Fortaleza, Ceará
  - CEDOES - Diagnóstico e Pesquisa, Vitória, Espírito Santo
  - Clínica SER da Bahia, Salvador, Estado de Bahia
  - L2IP - Instituto de Pesquisas Clínicas Ltda., Brasília, Federal District
  - IPC MT Instituto de Pesquisas Clinicas do Mato Grosso, Santo Ângelo, Mato Grosso
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - CMiP - Centro Mineiro de Pesquisa, Juiz de Fora, Minas Gerais
  - CETI - Centro de Estudos em Terapias Inovadoras Ltda., Curitiba, Paraná
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - LMK Serviços Médicos S/S Ltda, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, Sao Jose Rio Preto, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos - CEMEC, São Bernardo do Campo, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica e Serviços Médicos, São Paulo, São Paulo
  - A2Z Clinical Centro Avancado de Pesquisa Clinica, Valinhos, São Paulo
  - RDSS Ricardo Diaz Scientific Solution, São Paulo
- Bulgaria (7):
  - MC Artmed OOD, Plovdiv
  - UMHAT "Pulmed" OOD, Plovdiv
  - UMHAT-Plovdiv AD, Plovdiv
  - DCC 1 - Ruse, EOOD, Rousse
  - DCC 'Alexandrovska', EOOD, Sofia
  - DCC Focus 5 - MEOH OOD, Sofia
  - Military Medical Academy - MHAT - Sofia, Sofia
- Chile (5):
  - Centro Medico Prosalud, Santiago
  - CTR Estudios, Santiago
  - Enroll Spa, Santiago
  - BioMedica Research Group, Santiago
  - Clinical Research Chile SpA., Valdivia
- China (17):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Zhongshan TCM Hospital, Zhongshan, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Xiangya Hospital, Central South University, Changsha, Hu'nan
  - ZhuZhou Central Hospital, Zhuzhou, Hu'nan
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsushe
  - Jiujiang No.1 People's Hospital, Jiujiang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Province People's Hospital, Changchun, Jilin
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Renji Hospital Shanghai Jiaotong University School of Medicine - West Branch, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - The First Hospital of Jilin University, Changchun
- Colombia (8):
  - IPS Centro Medico Julian Coronel S.A., Cali, Valle del Cauca Department
  - Fundacion Cardiomet CEQUIN S.A.S, Armenia
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
  - Clínica de la Costa S.A.S, Barranquilla
  - Centro de Investigacion en Reumatologia y Especialidades Medicas CIREEM S.A.S., Bogotá
  - Servimed S.A.S., Bucaramanga
  - Preventive Care Ltda, Chía
  - Healthy Medical Center, Zipaquirá
- Czechia (2):
  - Revmatologie s.r.o., Brno
  - Fakultni nemocnice Olomouc, Olomouc
- CHU Clermont Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand, Drôme, France
- NNA Hospital, Athens, Attica, Greece
- Hungary (4):
  - Vita Verum Medical Egeszsegugyi Szolgaltato Bt., Székesfehérvár, Fejér
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Bekes Varmegyei Kozponti Korhaz, Gyula
  - Vital Medical Center, Veszprém
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Tel Aviv Sourasky Medical Center Pt, Tel Aviv
- Azienda Ospedaliera San Camillo Forlanini, Roma, Italy
- Japan (17):
  - JCHO Chukyo Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - NHO Chibahigashi National Hospital, Chiba, Chiba
  - KKR Hamanomachi Hospital, Fukuoka, Fukuoka
  - NHO Kyushu Medical Center, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu-shi, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Tonan Hospital, Sapporo, Hokkaido
  - Japanese Red Cross Society Himeji Hospital, Himeji-shi, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - NHO Yokohama Medical Center, Yokohama, Kanagawa
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo-To
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo-To
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku, Tokyo-To
- Mexico (10):
  - Clinica de Investigacion en Reumatologia y Obesidad S.C., Guadalajara, Jalisco
  - Centro de investigacion medica y reumatologia, Guadalajara, Jalisco
  - Centro de Investigacion Clínica GRAMEL S.C, Mexico City, Mexico City
  - Clinstile, S.A. de C.V., Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Dr. Salvador Zubiran, Mexico City, Mexico City
  - Consultorio Privado Dr. Miguel Cortes Hernandez, Cuernavaca, Morelos
  - Centro Peninsular de Investigacion Clinica, SCP, Mérida, Yucatán
  - Medical Care & Research SA de CV, Mérida, Yucatán
  - Investigacion y Biomedicina de Chihuahua, S.C., Chihuahua City
  - Centro de Investigacion y Atencion Integral Durango CIAID, Durango
- Peru (2):
  - Centro de Investigacion Clinica Inmunoreumatologia - ACQ Medic, Lima
  - HMA - Hospital Maria Auxiliadora, Lima
- Philippines (8):
  - Mary Mediatrix Medical Center, Lipa City, Batangas
  - Davao Doctors Hospital, Davao City, Davao Region
  - University of the Philippines Manila - Philippine General Hospital, Manila, National Capital Region
  - St. Luke's Medical Center, Quezon City, National Capital Region
  - Far Eastern University - Dr. Nicanor Reyes Medical Foundation, Quezon City, National Capital Region
  - Ospital Ng Makati, City of Taguig
  - The Medical City Iloilo, Iloilo City
  - Medical Center Manila, Manila
- Poland (7):
  - Nova Reuma Domysławska i Rusiłowicz, Spółka Partnerska Lekarza Reumatologa i Fizjoterapeuty, Bialystok
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Nzoz Bif-Med, Bytom
  - Pratia MCM Krakow, Krakow
  - Centrum Badawcze Panaceum Agnieszka Brzezicka, Magdalena Lenkiewicz Sp. z o.o., Malbork
  - Prywatna Praktyka Lekarska prof Pawel Hrycaj, Poznan
  - MICS Centrum Medyczne Warszawa, Warsaw
- Centro Reumatologico, Caguas, Puerto Rico
- Romania (4):
  - S.C Centrul Medical de Diagnostic si Tratament Ambulator Neomed S.R.L, Brasov
  - S C Delta Health Care SRL, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca
  - S.C.Centrul Medical Unirea SRL, Iași
- Serbia (3):
  - Institute of Rheumatology, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Clinical Center "Bezanijska Kosa ", Belgrade
- South Korea (2):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Hanyang University Seoul Hospital, Seoul
- Spain (4):
  - Hospital Universitario Marques de Valdecilla, Santander, Castellón
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Quironsalud Infanta Luisa, Seville
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan
- United Kingdom (2):
  - Guy's Hospital, London, Greater London
  - Doncaster Royal Infirmary, Doncaster, South Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/